CLINICAL TRIAL: NCT05463094
Title: A Randomized, Open-label, 2-Way-Crossover Study Assessing the Bioequivalence Between Single Doses of 500 mg Glucophage® XR RM Tablets (Merck/China Jiangsu-Manufactured) and 500 mg Glucophage® XR RM Tablets (Merck/Germany Darmstadt-Manufactured) Under Fed and Fasted State in Healthy Participants
Brief Title: GXR RM China BE Study (Darmstadt - Jiangsu)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200084_0030
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Glucophage® XR RM
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Test GXR RM (Fasted), Then Reference GXR RM (Fasted) (Experimental): Participants will receive a single dose of Test Glucophage Extended Release Reduced Mass (GXR RM) tablet on Day 1 in treatment period 1 followed by a single dose of Reference GXR RM tablet on Day 8 in treatment period 2 under fasted condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: Test Glucophage® XR; Drug: Reference Glucophage® XR
- First Reference GXR RM (Fasted), Then Test GXR RM (Fasted) (Experimental): Participants will receive a single dose of Reference GXR RM tablet on Day 1 in treatment period 1 followed by a single dose of Test GXR RM tablet on Day 8 in treatment period 2 under fasted condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: Test Glucophage® XR; Drug: Reference Glucophage® XR
- First Test GXR RM (Fed), Then Reference GXR RM (Fed) (Experimental): Participants will receive a single dose of Test GXR RM tablet on Day 1 in treatment period 1 followed by a single dose of Reference GXR RM tablet on Day 8 in treatment period 2 under fed condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: Test Glucophage® XR; Drug: Reference Glucophage® XR
- First Reference GXR RM (Fed), Then Test GXR RM (Fed) (Experimental): Participants will receive a single dose of Reference GXR RM tablet on Day 1 in treatment period 1 followed by a single dose of Test GXR RM tablet on Day 8 in treatment period 2 under fed condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: Test Glucophage® XR; Drug: Reference Glucophage® XR

INTERVENTIONS:
Drug: Test Glucophage® XR — Participants will receive single oral dose of Test GXR RM tablet under fasted or fed conditions.
  Other Names: Metformin hydrochloride
Drug: Reference Glucophage® XR — Participants will receive single oral dose of Reference GXR RM tablet under fasted or fed conditions.
  Other Names: Metformin hydrochloride

SUMMARY:
The purpose of this study is to assess Bioequivalence (BE), pharmacokinetics (PK), safety and tolerability following single oral dose administrations between a Glucophage Extended Release, Reduced Mass (Glucophage XR RM) manufactured in Merck Jiangsu China (test product) and that manufactured in Merck Darmstadt Germany (reference product) administered under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including medical history, ECG recording and physical examination judged by investigator.
* Participants with a body weight within 50 to 90 kg (kilogram) and BMI (body mass index) within the range 19 to 26 kg/m2 (kilogram per meter square).
* Participants with all values for biochemistry and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants with any surgical or medical condition, including findings in the medical history or in the pretrial assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation in the study or that could interfere with the study objectives, conduct or evaluation.
* Participants with history or presence of relevant liver diseases or hepatic or renal dysfunction.
* Participants with history of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility according to the Investigator's opinion.
* Participation in a clinical study within 90 days prior to first drug administration.
* Non-acceptance of study high-fat breakfast.
* Other protocol defined exclusion criteria could apply .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Metformin | Pre-dose up to 48 hours post-dose on Day 1 and Day 8
Maximum Observed Plasma Concentration (Cmax) of Metformin | Pre-dose up to 48 hours post-dose on Day 1 and Day 8

SECONDARY OUTCOMES:
Pharmacokinetic Plasma Concentrations of Metformin | Pre-dose up to 48 hours post-dose on Day 1 and Day 8
Number of Participants with Treatment-Emergent Adverse Events (AEs) | Baseline up to Day 10
Number of Participants with Abnormal Laboratory Variables, Vital Signs and 12-Lead Electrocardiogram (ECG) Measurements and Physical Examination | Baseline up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html